CLINICAL TRIAL: NCT04265469
Title: The Effect of Mobile Application in Foot Care of Type 2 Diabetes Patients: A Randomized Controlled Study
Brief Title: Mobile Application For Educating Diabetics About Foot Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Assistant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 42432568
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Foot, Mobile Application, Patient Education
Keywords: Diabetic foot, mobile application, patient education
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with diabetics get mobile education (Experimental): Patients with diabetics get mobile education
  Interventions: Other: Diabetic foot education
- Patients with diabetics (No Intervention): Patients with diabetics

INTERVENTIONS:
Other: Diabetic foot education — Give Diabetic foot education via mobile phone
  Arms: Patients with diabetics get mobile education

SUMMARY:
Purpose: Our aim was to develop a training program on the mobile application and to assess the effect of this training on the participants' knowledge about foot care, their self-efficacy and their behavior levels.

DETAILED DESCRIPTION:
The universe of this randomized controlled study consisted of 130 patients who had presented to a training and research hospital in Istanbul. The data were collected during the period March-September 2017 with an Information Form, the Diabetic Foot Knowledge Scale, Diabetic Foot Care Self-efficacy Scale, Foot Self-care Behavior Scale and a Feedback Form on the Mobile Application Training.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as a Type 2 diabetic according to ADA criteria at least six months prior to the study,
* being 18 years of age and over,
* being literate and fluent in Turkish,
* not having an active foot ulcer,
* owning and being able to operate a smart phone,
* not having any communication or mental problems,
* consenting to participating in the research.

Exclusion Criteria:

* Patients with advanced retinopathy and those wishing to withdraw from the research were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
their self-efficacy | change from baseline self efficiancy at week 4.
  Diabetic Foot Care Self-efficacy Scale is a scale that determines a diabetic individual's perception of self-efficacy with respect to executing diabetic foot care activities. Responses to this nine-item 10-point Likert-type of questionnaire are assessed on a visual scale that ranges from "I'm absolutely unsure=0" to "I'm very sure=10". The lowest possible score on the scale is 0; the highest is 100.
Diabetes Foot Knowledge | change from baseline Diabetes Foot Knowledge at week 4.
  Diabetes Foot Knowledge Questionnaire (DFKQ) were developed by Garcia et al. as a 5-item instrument that assesses the level of knowledge patients have about foot care. The questionnaire is evaluated on the basis of the total score. An increase in the score indicates that the diabetic individual has an increased level of knowledge about foot care
Foot Self-care Behavior | change from baseline Foot Self-care Behavior at week 4.
  Foot Self-care Behavior Scale assesses self-efficacy behavior in the context of foot care. It is a 16-item 5-point Likert-type of scale in which responses are assessed as "I do this: 1=Never, 2=Occasionally, 3=Sometimes, 4=Frequently, 5=Always." The lowest possible score on the scale is 16; the highest is 80